CLINICAL TRIAL: NCT05008523
Title: Evaluation of an Experimental Educational Module on Opioid-related Occupational Safety to Minimize Barriers toOverdose Response Among Police Officers
Brief Title: Opioids and Police Safety Study
Acronym: OPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY2019-3315
Record Dates: First submitted 2021-06-21; First posted 2021-08-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-03

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose | interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: The Opioids and Police Safety Study employed a pragmatic trial design evaluated in a simultaneous embedded mixed-method approach.
Masking Description: Participants are randomized to the experimental or the control arm for occupational risk reduction trainings. Trainings are not designated as experimental or control.
  CHANGE TO PROTOCOL: Control dropped to enable recruitment. Outcome measures are the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioids and Police Safety Occupational Risk Reduction Training (Experimental): Provides occupational risk reduction training for police in 49 slides including 8 filmed videos (police officers, MDs, SSP staff, a person in recovery). The training is delivered online with secure access only for enrolled study participants.
  Interventions: Behavioral: Opioids and Police Safety Occupational Risk Reduction Training (OPS)
- COVID Occupational Risk Reduction Training (Active Comparator): The COVID-19 and Police Safety training (Control only) includes 22 slides, also narrated by a professional voice narrator.
  Interventions: Behavioral: Opioids and Police Safety Occupational Risk Reduction Training (COVID)

INTERVENTIONS:
Behavioral: Opioids and Police Safety Occupational Risk Reduction Training (OPS) — Potential participants are provided with a flyer with directions to enroll online. Groups are randomized by zip code (all participants with the same zip code receive the same training to avoid contamination by precinct) Both the experimental and control groups first take the online GetNaloxoneNow.org First Responder training; then the experimental group takes the online OPS training and the control group takes the online COVID training. Both groups take a pre-survey prior to both trainings and a post-survey after they complete both trainings. Both groups also receive (via email) a resource list with information that was provided in their respective trainings plus additional resources re: occupational risk reduction appropriate to each training. Every quarter for one year, participants are emailed a reminder to get back online to take the survey again.
  Other Names: OPS
  Arms: Opioids and Police Safety Occupational Risk Reduction Training
Behavioral: Opioids and Police Safety Occupational Risk Reduction Training (COVID) — Potential participants are provided with a flyer with directions to enroll online. Groups are randomized by zip code (all participants with the same zip code receive the same training to avoid contamination by precinct) Both the experimental and control groups first take the online GetNaloxoneNow.org First Responder training; then the experimental group takes the online OPS training and the control group takes the online COVID training. Both groups take a pre-survey prior to both trainings and a post-survey after they complete both trainings. Both groups also receive (via email) a resource list with information that was provided in their respective trainings plus additional resources re: occupational risk reduction appropriate to each training. Every quarter for one year, participants are emailed a reminder to get back online to take the survey again.
  Other Names: COVID
  Arms: COVID Occupational Risk Reduction Training

SUMMARY:
Overdose deaths are currently the largest cause of accidental death in the US and opioid-related overdose deaths constitute the overwhelming majority of these deaths. Demands for a knowledge-base for effective law enforcement interventions is growing. This proposed study is designed to provide a knowledge base regarding key obstacles and facilitators of the willingness and preparedness of police to administer naloxone and related risk reduction practices and evaluate the efficacy of a web-based opioid-related occupational safety and risk reduction curriculum. Findings from this study will be applied to the development and implementation of effective interventions for police officers aimed at harmonizing law enforcement practices with public health goals.

DETAILED DESCRIPTION:
This application proposes to contribute to the harmonization of law enforcement practices and public health goals to combat rising morbidity and mortality rates associated with opioid-related overdose (OD). Police departments around the U.S. are increasingly making the OD reversal drug, naloxone, available to their officers. This intervention has the potential to greatly improve emergency response after an OD. The proportion of precincts mandating that officers carry naloxone remains small, however, and barriers remain that make adoption of these first-responder programs problematic. Lawsuits from police unions contesting naloxone- related mandates and occupational safety concerns, including the potential for needle stick injuries (HIV/HCV risk) and incidental contact with fentanyl-class substances, constitute barriers, as do stigma and concerns about legal jeopardy. The study team proposes to equip police with best-practices for minimizing workplace harms related to encounters with PWUO/PWID and the legal and practical knowledge to respond confidently to an OD without fear of legal jeopardy as well as reduce health risks to PWUOs and PWIDs associated with law enforcement. More than 10,000 law enforcement officers in Pennsylvania (roughly one third of all PA officers) have already received naloxone and OD response training from GetNaloxoneNow.org (GNN), a web-based intervention. With the support of county departments of health, harm reduction agencies, law enforcement, and district attorneys, the team proposes to adapt extant interventions for police to create an online training module aimed at reducing barriers to police engagement in OD response. Using a mixed-method design, organized around a pragmatic trial design, the study will achieve the following objectives:1) Adapt an occupational risk reduction (ORR) curriculum to add to a web-based OD response and naloxone training platform (GNN); 2) Describe naloxone use patterns, OD response experiences, and attitudes related to illicit opioid use among a sample (N = 300) of police officers in PA trained via the GNN platform; 3) Evaluate the relative effectiveness of ORR + GNN, compared with GNN-only, with respect to the following outcomes: a) rates of carrying naloxone while on/off-duty; b) rates of OD response in which naloxone is/isn't administered; c) numbers of referrals to treatment; d) numbers of syringes confiscated; and e) rates of information sharing with OD survivors and others. Mediators and moderators of efficacy will also be analyzed. 4) Document the range of psychosocial mechanisms underlying participant OD response engagement post-intervention. This study aims to remove barriers to life-saving police engagement with PWUO/PWID by focusing both on the safety of law enforcement and evidence-based and best-practices for working with persons at risk of an opioid OD. The study also will provide empirical evaluation of the diffusion of naloxone-based response among law enforcement.

ELIGIBILITY:
Inclusion Criteria:

* Active duty Police Officer

Exclusion Criteria:

* Desk only- not active duty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Naloxone Behavioral Outcomes in Policing Procedure | Time frame for all above items: the past 30 days at the time the survey is being administered; [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Number of days during the past 30 days in which participants had naloxone available and carried naloxone while at work.
Change in Naloxone Behavioral Outcomes in Policing Procedure | Time frame for all above items: the past 30 days at the time the survey is being administered; [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Number of days during the past 30 days in which participants had naloxone available and carried naloxone outside of work hours.
Change in Naloxone Behavioral Outcomes in Policing Procedure | Time frame for all above items: the past 30 days at the time the survey is being administered; [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Number of days during the past 30 days in which participants responded to an OD event, attempted to intervene, and/or administered naloxone.
Change in Referral Behavioral Outcomes in Policing Procedure | Time frame: the past 30 days at the time the survey is being administered; [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Number of referrals to evidence-based or other drug treatment or social services made during the past 30 days.
Change in Confiscation Behavioral Outcomes in Policing Procedure | Time frame for all above items: the past 30 days at the time the survey is being administered; [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Number of episodes involving syringe confiscation in the past 30 days (with/without proper technique).
Change in Confiscation Behavioral Outcomes in Policing Procedure | Time frame for all above items: the past 30 days at the time the survey is being administered; [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Number of episodes in the past 30 days involving drug confiscation (with/without proper technique).

SECONDARY OUTCOMES:
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Which of the following diseases is MOST likely to be transmitted by a needle stick injury?
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  The risk of getting a bloodborne infection as a result of a needle stick injury is high (check only one response).
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  To avoid being stuck with a needle, police officers should (select ALL that apply)
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  The evidentiary value of syringes and any drug residue therein is (fill in the blank by checking only one response).
  5) Possession of syringes is (fill in the blank by checking only one response). 6) Confiscating syringes from people who inject drugs... (check all that apply): 7) Testing and precautionary treatment of any NSI is important, because... (fill in the blank by checking only one response).
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Possession of syringes is (fill in the blank by checking only one response). 6) Confiscating syringes from people who inject drugs... (check all that apply): 7) Testing and precautionary treatment of any NSI is important, because... (fill in the blank by checking only one response).
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Confiscating syringes from people who inject drugs... (check all that apply):
  7) Testing and precautionary treatment of any NSI is important, because... (fill in the blank by checking only one response).
Change in participant knowledge about needle stick injury and treatment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Testing and precautionary treatment of any NSI is important, because... (fill in the blank by checking only one response).
Degree of participant familiarity with proper technique for dealing with contaminated injection equipment | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Please indicate your agreement with the following statements relating to needle stick prevention and response (1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree):
  1. I feel confident in my ability to avoid needlestick injuries.
  2. I feel confident in my ability to get people who inject drugs to tell me if they have sharps before I search them.
  3. I feel confident in my ability to conduct a Terry Stop with minimal risk of a needlestick injury.
  4. In the event of needle stick injury, I would know the response protocol.
  5. In the event of a needle stick injury, I feel confident in my ability to get the right testing and medical care.
  6. In the event of a needle stick injury, I feel comfortable talking to the owner of the needle about coming with me to get tested.
Degree of participant awareness of post-exposure prophylaxis (PEP) and its uses | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  (1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree):
  1. A first responder's risk of experiencing an overdose from touching fentanyl is high (select one response)
  2. A first responder's risk of experiencing an overdose from breathing fentanyl is high (select one response)
  3. Possession of naloxone by civilians is authorized only when accompanied with a valid prescription (select one response)
  4. The 911 Good Samaritan Law... (fill in the blank and select all that apply)
  5. When called to an overdose scene, it is best practice for police officers to... (fill in the blank and select all that apply)
Degree of participant awareness of risk of fentanyl exposure and proper technique for dealing with synthetic opioids | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Response options: (1 = all the time, 2 = most of the time, 3 = sometimes, 4 = rarely, 5 = never):
  1. I am confident that I won't overdose from incidental skin contact with fentanyl.
  2. I am confident about my ability to use basic protective equipment to avoid fentanyl exposure.
  3. I am confident that I can recognize an opioid overdose when I see it.
  4. I am confident that I can effectively reverse an overdose using rescue techniques and naloxone.
  5. I am confident that I know how to conduct myself at an overdose scene to safeguard public health and public safety.

OTHER OUTCOMES:
Degree of participant familiarity with fentanyl-class substances | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  * Over your career, how often have you been exposed to touching or breathing in powder fentanyl?
  * A first responder's risk of experiencing an overdose from touching fentanyl is high
  * A first responder's risk of experiencing an overdose from breathing fentanyl is high Response options: 1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree)
Degree of participant familiarity with best-practices related to policing PWUO and PWID who may be carrying heroin contaminated with fentanyl-class substances | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  * I am confident that I won't overdose from incidental skin contact with fentanyl.
  * I am confident about my ability to use basic protective equipment to avoid fentanyl exposure Response options: 1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree
Opioid-Related OD knowledge | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  The items related to a participant's ability to recognize and respond to an opioid-related overdose, with or without naloxone, were adapted from the Opioid Overdose Knowledge Scale (OOKS).
  * I am confident that I can effectively reverse an overdose using rescue techniques and naloxone
  * I am confident that I can recognize an opioid overdose when I see it.
  * I am confident that I know how to conduct myself at an overdose scene to safeguard public health and public safety Response options: 1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree
Hypothesized Mediators of Intervention Efficacy: Stigma | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Response options: 1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree Providing naloxone to people with addiction enables more risky drug use Distributing naloxone widely in the community is a good way to reduce overdose fatalities Rapidly giving a lot of naloxone (blasting) when reversing an overdose is a good way to teach someone a lesson It is important to prevent overdose risk directly following a period of incarceration I worry about my safety when I encounter people with addiction People with addiction make communities less safe People with addiction can make positive health choices to protect themselves or others When people with addiction are placed in secure /mandated treatment facilities, communities are better off A lot of people with addiction are outsiders coming into communities to peddle drugs
Potential Moderators: Demographic Variables | Baseline
  1. Age This construct will be assessed via the following item: What is your age (in years)?
  2. Sex This construct will be assessed via the following multiple choice item: What is your gender?
  3. Law enforcement rank This construct will be assessed via the following multiple choice item: What is your current rank?
  4. Number of years on the job This construct will be assessed via the following item: What is the total number of years you have been working in law enforcement (including work in PA and other states, if relevant)?
Potential Moderators: Perceived Attitudes/Expectations | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Response options: 1 = strongly agree, 2 = agree, 3 = neither agree nor disagree, 4 = disagree, 5 = strongly disagree
  1. My police agency values administering naloxone.
  2. My police agency values linking people who use drugs to treatment.
  3. My department does not appreciate effort from me to help people who use drugs get treatment and stay alive.
  4. My agency would ignore any complaint from me regarding officer misconduct toward people who use drugs.
  5. The agency cares that I do not get hurt by needlestick injuries.
  6. The agency is willing to extend itself in order to help me stay safe when handling needles.
  7. Helping people who are addicted to drugs is a part of determining who gets promoted in my police agency.
  8. The agency cares about my opinions about people who use drugs.
  9. The agency wishes to give me all the available resources possible for helping people who use drugs.
Prior instances of witnessing an opioid-related overdose | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  The following questions relate to your experiences with opioid overdose. For each item, please choose what best describes your response to each statement (select ONLY one for each item).
  1. Over your career, how often have you been at the scene of overdose emergencies?
  2. Over your career, how often have you administered naloxone to a civilian experiencing an overdose?
  3. Over your career, how often have you administered naloxone to a law enforcement officer experiencing an overdose?
  4. Over your career, how often have you been exposed to touching or breathing in powder fentanyl?
Prior instances of working with syringes | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  The following questions cover your experiences with syringes in the line of duty. Select the one best response for each item:
  1. In the last 3 months, how often have you transported syringes (for evidence or other reasons)?
  2. In the last 3 months, how often have you discarded syringes in the trash?
  3. In the last 3 months, how often have you confiscated syringes from an individual?
  4. In the last 3 months, how often have you confiscated naloxone/Narcan?
  5. In the last 3 months, how often have you arrested someone for syringe possession?
  6. In the last 3 months, how often have you arrested someone for drug possession?
  7. Over your entire policing career, how often have you been accidentally stuck by a needle?
  8. In the last 3 months, how often were you accidentally stuck by a needle?
  9. In the last 3 months, how often have you been at scenes of overdoses?
Prior instances responding to an overdose | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  Now please tell us just about the following events which you may have experienced when responding to an overdose in the past 3 months.
  1. When responding to ODs in the past 3 months, how often were you or your partner exposed to fentanyl class drugs?
  2. When responding to ODs in the past 3 months, how often have you informed someone about the 911 Good Samaritan Law?
  3. When responding to ODs in the past 3 months, how often have you arrested someone at the scene?
  4. When responding to ODs in the past 3 months, how often have you administered naloxone to a civilian?
Experiences with other programs | [Data collected: Baseline, Post Intervention: 90 days, 180 days, 270 days, 360 days]
  This next set of questions relate to your experiences with other programs in addressing the overdose crisis in your community:
  1. In the last 3 months, how often have you provided information about or made referrals to drug treatment programs?
  2. In the last 3 months, how often have you made referrals to syringe service programs?
  3. In the last 3 months, how often have you made referrals to naloxone distribution programs?
  4. In the last 3 months, how often have you made referrals to social support (e.g. housing, employment) programs?

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simmons J, Elliott L, Bennett AS, Beletsky L, Rajan S, Anders B, Dastparvardeh N. Evaluation of an Experimental Web-based Educational Module on Opioid-related Occupational Safety Among Police Officers: Protocol for a Randomized Pragmatic Trial to Minimize Barriers to Overdose Response. JMIR Res Protoc. 2022 Feb 25;11(2):e33451. doi: 10.2196/33451. PMID 35212639

DOCUMENTS (1):
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT05008523/ICF_000.pdf